CLINICAL TRIAL: NCT05095987
Title: Evaluation of One Day Discharge After Laparoscopic Appendectomy for Uncomplicated Appendicitis in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miro Jukić (Other)
Responsible Party: Sponsor-Investigator, Miro Jukić, MD, PhD, attending Pediatric Surgeon, University Hospital of Split
Organization: University Hospital of Split (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHSplitpedsurg
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Appendicitis Acute
Keywords: Pediatric Surgery; One day discharge; parental satisfaction questionnaire; laparoscopic appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: prospective nonrandomized cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One day discharge after laparoscopic Appendectomy (Experimental)
  Interventions: Procedure: Laparoscopic Appendectomy

INTERVENTIONS:
Procedure: Laparoscopic Appendectomy — Laparoscopic Appendectomy for acute uncomplicated appendicitis in children

SUMMARY:
The aim of this study was to evaluate the value and safety of discharge of a child to home care within 24 hours after laparoscopic appendectomy for uncomplicated appendicitis to reduce the impact on the child's psyche and need for hospitalisation. Baseline demographic data and intraoperative finding will be recorded. Parents are given a two-page questionnaire that is completed in three cycles (immediately after discharge, daily until the first control and immediately before the first control). All data will be statistically processed using descriptive statistics.

DETAILED DESCRIPTION:
The research would include children who underwent laparoscopic surgery due to uncomplicated acute appendicitis in the period from October 2021 to October 2023 at the Clinic for Pediatric Surgery of the University Hospital Center Split. After the suspicion of acute inflammation of the appendix is established, the pediatric surgeon decides on surgical treatment. Recently, laparoscopic appendectomy has been performed in a standardized manner at the Clinic for Pediatric Surgery of the Clinical Hospital Center Split. After the operation, and in the current practice, the children would stay in hospital for 2 to 4 days. As the generally known psychological aspects of changes in children's behaviour in involuntary hospital stays, and now even more pronounced due to the SARS-CoV-2 (Severe acute respiratory syndrome coronavirus 2) COVID19 virus pandemic and reduced opportunities for parents to stay with children, the main goal of this study is to evaluate and possibly reduce hospital stay to a minimum and proof that there are no complications in treatment outcomes due to shortening the length of hospital treatment. To conduct this research, parents are given a two-page questionnaire that is completed in three cycles (immediately after discharge, daily until the first control and immediately before the first control). Baseline demographic data and intraoperative findings will be recorded. All data will be statistically processed using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* children 6 to 18 years
* uncomplicated acute appendicitis treated with laparoscopic approach
* children released within 24 hours

Exclusion Criteria:

* children under 6 years
* complicated acute appendicitis
* intraoperative complication
* operated by classical approach
* children needing longer hospital care and parental therapy
* children with significant comorbidities that could affect treatment outcomes

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Safety of one day discharge after laparoscopic Appendectomy | 4 weeks
  Safety of one day discharge after laparoscopic appendectomy for uncomplicated acute appendicitis in children.
  It will be measured by readmission rate of the "early" discharged children (within 24 hours from surgery). If there is no readmissions then the one day discharge after laparoscopic appendectomy for uncomplicated acute appendicitis in children would be considered safe. Again, the condition of an operated child is monitored and followed-up in an outpatient clinic 1 week after the surgery. The parental notes, and observations are taken into account.

SECONDARY OUTCOMES:
Parental Satisfaction | 1 week
  Using a questionnaire to evaluate parental satisfaction. There are four parts of the questionnaire: First part of the questionnaire 3 level scoring in satisfaction in agreeing of one day discharge after the surgery (the very first day), second part is structured as a simple yes/no answer possibility of childs behaviour and pain at home. The third part is a child pain score from 0-10, 0 being no pain and 10 greatest unbearable pain and parental-child pain management (used medicine, etc...). Finally, fourth part is modified first part where there is 3 level scoring in satisfaction in agreeing of one day discharge after the surgery, but now one week after.

OTHER OUTCOMES:
Readmission rate | 2 weeks
  Readmission rate to the hospital due to the laparoscopic appendectomy.
Complication rate | 2 weeks
  Complication due to surgical intervention
Cost reduction | 2 weeks
  due to shorter hospital stay the study anticipates a cost reduction

CONTACTS AND LOCATIONS:
Overall Officials: Miro Jukić, MD, PHD, Study Director — University Hospital of Split
Locations (1):
- University hospital of Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT05095987/Prot_SAP_000.pdf